CLINICAL TRIAL: NCT04510480
Title: Systems Saving Lives - Long-term Survival of Out-of-hospital Cardiac Arrest in the Urban Area of Bologna Following the Implementation of the Pre-arrival Instructions, the DAE RespondER, Mechanical Chest Compressors and Circulatory Support With REBOA and ECMO
Brief Title: Systems Saving Lives - Long-term Survival of Out-of-hospital Cardiac Arrest in the Urban Area of Bologna
Acronym: SSL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1.0
Record Dates: First submitted 2020-07-09; First posted 2020-08-12 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cardiac arrest: Out of hospital cardiac arrest patients (Historical cohort) from 1st January 2009 and 30th June 2020.
  Out of hospital cardiac arrest patients from 1st July 2020 and 31st December 2025.
  Interventions: Other: Observational study without specific intervention

INTERVENTIONS:
Other: Observational study without specific intervention — Observational study with standard cardiac arrest approach

SUMMARY:
Evaluation of clinical, logistical, and technical factors (e.g. implementation of pre-arrival instructions, implementation of the DAE RespondER, mechanical chest compressor, REBOA, and E-CPR) that impact on the outcomes of out-of-hospital cardiac arrest patients.

ELIGIBILITY:
Inclusion Criteria:

* Out of Hospital cardiac arrest patients (historical cohort) from 1st January 2009 and 30th June 2020
* Out of Hospital cardiac arrest patients from 1st July 2020 and 31st December 2025

Exclusion Criteria:

* False cardiac arrest
* In-hospital cardiac arrest

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population served by EMS of Bologna area
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ROSC (Return of spontaneous circulation) | 1st July 2020 to 31st December 2025
  ROSC (Return of spontaneous circulation) of cardiac arrest patients
Hospital admission status | 1st July 2020 to 31st December 2025
  Hospital admission status of cardiac arrest patients
Hospital discharge status/survival at 30 days | 30 days
  Hospital discharge status/survival at 30 days of cardiac arrest patients

SECONDARY OUTCOMES:
Survival at 6 months | 6 months
  Survival at 6 months of cardiac arrest patients
Survival at 1 years | 1 year
  Survival at 1 years of cardiac arrest patients

CONTACTS AND LOCATIONS:
Overall Officials: Federico F Semeraro, MD, FERC, Principal Investigator — Maggiore Hospital Carlo Alberto Pizzardi AUSL di Bologna
Locations (1):
- Maggiore Hospital Ospedale Maggiore Carlo Alberto Pizzardi AUSL di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grasner JT, Wnent J, Herlitz J, Perkins GD, Lefering R, Tjelmeland I, Koster RW, Masterson S, Rossell-Ortiz F, Maurer H, Bottiger BW, Moertl M, Mols P, Alihodzic H, Hadzibegovic I, Ioannides M, Truhlar A, Wissenberg M, Salo A, Escutnaire J, Nikolaou N, Nagy E, Jonsson BS, Wright P, Semeraro F, Clarens C, Beesems S, Cebula G, Correia VH, Cimpoesu D, Raffay V, Trenkler S, Markota A, Stromsoe A, Burkart R, Booth S, Bossaert L. Survival after out-of-hospital cardiac arrest in Europe - Results of the EuReCa TWO study. Resuscitation. 2020 Mar 1;148:218-226. doi: 10.1016/j.resuscitation.2019.12.042. Epub 2020 Feb 3. PMID 32027980
- [Result] Grasner JT, Lefering R, Koster RW, Masterson S, Bottiger BW, Herlitz J, Wnent J, Tjelmeland IB, Ortiz FR, Maurer H, Baubin M, Mols P, Hadzibegovic I, Ioannides M, Skulec R, Wissenberg M, Salo A, Hubert H, Nikolaou NI, Loczi G, Svavarsdottir H, Semeraro F, Wright PJ, Clarens C, Pijls R, Cebula G, Correia VG, Cimpoesu D, Raffay V, Trenkler S, Markota A, Stromsoe A, Burkart R, Perkins GD, Bossaert LL; EuReCa ONE Collaborators. EuReCa ONE-27 Nations, ONE Europe, ONE Registry: A prospective one month analysis of out-of-hospital cardiac arrest outcomes in 27 countries in Europe. Resuscitation. 2016 Aug;105:188-95. doi: 10.1016/j.resuscitation.2016.06.004. Epub 2016 Jun 16. PMID 27321577
- [Result] Del Giudice D, Semeraro F, Ristagno G, Picoco C, Cordenons F, Dell'Arciprete O, Mora F, Scapigliati A, Gordini G. DAE RespondER: The Emilia Romagna app for a regional "community saving lives" system. Resuscitation. 2019 Dec;145:34-36. doi: 10.1016/j.resuscitation.2019.10.002. Epub 2019 Oct 15. No abstract available. PMID 31626865
- [Result] Oving I, Masterson S, Tjelmeland IBM, Jonsson M, Semeraro F, Ringh M, Truhlar A, Cimpoesu D, Folke F, Beesems SG, Koster RW, Tan HL, Blom MT; ESCAPE-NET Investigators. First-response treatment after out-of-hospital cardiac arrest: a survey of current practices across 29 countries in Europe. Scand J Trauma Resusc Emerg Med. 2019 Dec 16;27(1):112. doi: 10.1186/s13049-019-0689-0. PMID 31842928
- [Result] Di Marco S, Tucci R, Tonelli G, Frione G, Semeraro F, Ristagno G, Scapigliati A. Preparedness for telephone dispatch-assisted cardiopulmonary resuscitation in Italy. A National survey. Resuscitation. 2020 Apr;149:87-88. doi: 10.1016/j.resuscitation.2020.02.007. Epub 2020 Feb 18. No abstract available. PMID 32084569
- [Result] Semeraro F, Gamberini L, Tartaglione M, Mora F, Dell'Arciprete O, Cordenons F, Del Giudice D, Picoco C, Gordini G. An integrated response to the impact of coronavirus outbreak on the Emergency Medical Services of Emilia Romagna. Resuscitation. 2020 Jun;151:1-2. doi: 10.1016/j.resuscitation.2020.03.005. Epub 2020 Mar 20. No abstract available. PMID 32205158
- [Result] Scquizzato T, Burkart R, Greif R, Monsieurs KG, Ristagno G, Scapigliati A, Semeraro F. Mobile phone systems to alert citizens as first responders and to locate automated external defibrillators: A European survey. Resuscitation. 2020 Jun;151:39-42. doi: 10.1016/j.resuscitation.2020.03.009. Epub 2020 Apr 3. No abstract available. PMID 32251700
- [Result] Nolan JP, Monsieurs KG, Bossaert L, Bottiger BW, Greif R, Lott C, Madar J, Olasveengen TM, Roehr CC, Semeraro F, Soar J, Van de Voorde P, Zideman DA, Perkins GD; European Resuscitation Council COVID-Guideline Writing Groups. European Resuscitation Council COVID-19 guidelines executive summary. Resuscitation. 2020 Aug;153:45-55. doi: 10.1016/j.resuscitation.2020.06.001. Epub 2020 Jun 7. PMID 32525022
- See also: EMS regional website — https://www.118er.it/
- See also: DAE RespondER website — https://www.118er.it/dae/